CLINICAL TRIAL: NCT06549101
Title: Neutrophil-to-Lymphocyte Ratio and Mortality After Emergency Surgery
Brief Title: NLR and Emergency Surgery
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Other Study IDs: OAIC 37/22
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-08

CONDITIONS: Emergency Surgery
Keywords: Neutrophil-to-lymphocyte ratio; Emergency surgery; NLR

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In the immune system, it has been observed that the preoperative neutrophil-to-lymphocyte ratio (NLR) is an index that reflects the state of inflammation and oxidative stress. In the perioperative period, NLR has been described as a predictor for patients who will develop renal injury, ischemic stroke, and myocardial injury. Since preoperative inflammation is a predictor of morbidity and mortality in patients undergoing non-cardiac surgery, a retrospective analysis of the inflammatory status of patients undergoing surgery at the center is proposed.

DETAILED DESCRIPTION:
A retrospective analysis of patients operated on at the Clinical Hospital of the University of Chile is proposed. The search will be conducted in the electronic medical records of all patients operated on between January and December 2021, with no exclusion criteria for this analysis. Demographic data, complications, length of hospital stay, and specific characteristics such as the need for mechanical ventilation, time spent in intermediate care units, and ICU as well as total hospitalization time will be recorded. For the purpose of this study, the preoperative complete blood count of the patients will be analyzed to search for hematological variables that reflect the state of preoperative systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Availability of complete blood count in electronic medical records of all patients operated on between January and December 2021

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Emergency patients operated on at the Clinical Hospital of the University of Chile between January and December 2021
Sampling Method: Non-Probability Sample
Enrollment: 851 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
NLR | Day of surgery
  Preoperative neutrophil-to-lymphocyte ratio
Mortality | 6 months after surgery
  30 and 180 days mortality

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Maldonado, M.D., M. Sc., Study Chair — Hospital Clínico de la Universidad de Chile
Locations (1):
- Hospital Clínico de la Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maldonado F, Albornoz M, Enriquez I, Espinoza C, Chang H, Carrasco L, Diaz-Papapietro C, Medina F, Gonzalez R, Caceres M. Association of neutrophil-to-lymphocyte ratio with age and 180-day mortality after emergency surgery. BMC Anesthesiol. 2024 Sep 17;24(1):329. doi: 10.1186/s12871-024-02718-z. PMID 39289610